CLINICAL TRIAL: NCT00232661
Title: A Randomised, Double-blind, Study Comparing ARIMIDEX™ With NOLVADEX™ as Neo-adjuvant and Adjuvant Treatment in Post-menopausal Women With Large Operable (T2 (≥3cm), T3, N0-2, M0) or Potentially-operable, Locally Advanced (T4b, N0-2, M0), ER+ and/or PR+ Breast Cancer.
Brief Title: PROACT - Pre-Operative Arimidex Compared To Tamoxifen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Francisco Sapunar, MD - Arimidex Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1033IL/0039; D5395C00039
Record Dates: First submitted 2005-09-30; First posted 2005-10-05 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: ARIMIDEX (anastrazole)
Drug: NOLVADEX (tamoxifen)

SUMMARY:
The purpose of this study is to compare tamoxifen, versus a newer treatment, ARIMIDEX, which we already know to be well tolerated. The main objectives of this research study are to see whether using these drugs will shrink down tumours before surgery and to see if any shrinkage in the tumour affects the extent of surgery that is required.

ELIGIBILITY:
Inclusion Criteria:

* Operable or potentially operable breast cancer
* Invasive breast cancer proven to be hormone-sensitive (ER+/PR+)
* Patients who might benefit from endocrine treatment prior to surgery
* Postmenopausal
* Signed written informed consent

Exclusion Criteria:

* Inoperable breast cancer
* Patient unwilling to undergo surgery
* Any reason why the patient may not be able to conform to study requirements
* Any previous treatment for breast cancer
* Previous Tamoxifen use as a part of breast cancer prevention trials
* Not willing to stop taking drugs that affect sex-hormones such as HRT
* Previous history of breast cancer
* Previous history of invasive malignancy within the last 10 years
* Any other severe disease that may prevent surgery, place the patient at risk, or influence the study results
* Treatment with an experimental drug within the last 3 months
* Risk of transmitting HIV, Hepatitis B or C

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2000-08; Primary Completion 2003-01 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Objective tumour response | Assessed at 3 months

SECONDARY OUTCOMES:
Pathological response | Assessed at 3 months
Extent of breast surgery | Assessed at 3 months
Extent of axillary down-staging | Assessed at 3 months
Clinical ultrasound response versus clinical caliper response | Assessed at 3 months
Safety | Assessed up to 5 years + 30 days
Complications due to surgery | Assessed up to 30 days post-surgery
Health economics outcomes | Assessed up to 30 days post-surgery
Quality of Life assessments | Assessed at 3 months
Effect of ethnicity with respect to baseline patient and tumour characteristics, safety and objective tumour response rate | Assessed up to 5 years + 30 days
Recurrence-free survival and survival | Assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Arimidex Medical Science Director, MD, Study Director — AstraZeneca
Locations (79):
- United States (13):
  - Research Site, Santa Rosa, California
  - Research Site, New Britain, Connecticut
  - Research Site, Torrington, Connecticut
  - Research Site, Springfield, Illinois
  - Research Site, Mason City, Iowa
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Pittsfield, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, Portland, Oregon
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Olympia, Washington
- Belgium (4):
  - Research Site, Antwerp
  - Research Site, Hasselt
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (6):
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo, São Paulo
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Sheffield
- Canada (5):
  - Research Site, Edmonton, Alberta
  - Research Site, Newmarket, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Czechia (6):
  - Research Site, Brno
  - Research Site, Nová Ves pod Pleší
  - Research Site, Olomouc
  - Research Site, Peské Budjovice
  - Research Site, Prague
  - Research Site, Praha-5
- France (10):
  - Research Site, Lyon, Cedex 08
  - Research Site, Avignon
  - Research Site, Dijon
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Tours
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Szeged
  - Research Site, Szolnok
- Italy (8):
  - Research Site, Bologna, BO
  - Research Site, Cagliari, CA
  - Research Site, Monserrato, CA
  - Research Site, Kashiwa, Chiba
  - Research Site, Florence, FI
  - Research Site, Genova, GE
  - Research Site, Palermo, PA
  - Research Site, Reggio Emilia, RE
- Japan (19):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Chiba, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyushu, Fukuoka
  - Research Site, Ōta, Gunma
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Amagasaki, Hyōgo
  - Research Site, Isehara, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Niigata, Niigata
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Osaka, Osaka
  - Research Site, Sayama, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Kitaadachi, Saitama
  - Research Site, Chūō, Tokyo
- Netherlands (3):
  - Research Site, Nijmegen
  - Research Site, Sittard
  - Research Site, The Hague

REFERENCES:
- [Result] Cataliotti L, Buzdar AU, Noguchi S, Bines J, Takatsuka Y, Petrakova K, Dube P, de Oliveira CT. Comparison of anastrozole versus tamoxifen as preoperative therapy in postmenopausal women with hormone receptor-positive breast cancer: the Pre-Operative "Arimidex" Compared to Tamoxifen (PROACT) trial. Cancer. 2006 May 15;106(10):2095-103. doi: 10.1002/cncr.21872. PMID 16598749
- [Derived] Fujiwara Y, Takatsuka Y, Imoto S, Inaji H, Ikeda T, Akiyama F, Tamura M, Miyoshi K, Iwata H, Mitsuyama S, Noguchi S. Outcomes of Japanese breast cancer patients treated with pre-operative and post-operative anastrozole or tamoxifen. Cancer Sci. 2012 Mar;103(3):491-6. doi: 10.1111/j.1349-7006.2011.02171.x. Epub 2012 Jan 13. PMID 22136317